CLINICAL TRIAL: NCT04973553
Title: Finding the Optimal Session Length of Upper Limb Rehabilitation of People With Moderate to Severe Upper Limb Sensorimotor Impairments After Acute Stroke: A Dose Escalation Study
Brief Title: Dose Escalation Upper Limb Rehabilitation in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOMINO-001
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants with acute stroke (Experimental): (a) a first-ever unilateral, diagnosed stroke by a neurologist as defined by the World Health Organisation, (b) been admitted to the acute hospital for rehabilitation, (c) Upper limb hemiparesis or hemiplegia with a trace of muscle contraction:≥grade 1 at shoulder (abductors or elevators) or wrist/finger extensors measured by the MRC Scale and a score of <61 on the Motricity Index and severely motor affected by score of 2 or 3 on item number 5 on the NIH Stroke Scale (NIHSS)[24], (d) the age of > 18 years and (e) the ability to provide informed consent.
  Interventions: Other: upper limb rehabilitation

INTERVENTIONS:
Other: upper limb rehabilitation — the intervention consisting of two components: a) Upper limb training protocol; b) Technology-assist training.

SUMMARY:
A phase 1, single-ascending dose clinical trial will be conducted. This study will be designed to test increasing doses of multimodal exercise in successive cohorts of six participants (cumulative 3 + 3 design)[22] (Figure 1).

Maximum dose is reached when two or more participants experience DLT. DLT, dose-limiting tolerance.

The 'dose' will be defined as the ability to reach a fixed maximal level of exercise (type, duration (including session length) in the first two weeks post-stroke without experiencing dose-limiting tolerance (DLT). DLT thresholds will be based on failure to completeshould be less than 80% of prescribed 3-day rehabilitation dose due to pain, rate of perceived exertion, fatigue, or effort required.

Rehabilitation and measurement sessions will be held at either at the Stroke or Geriatric Units at Campus Sint-Jan, Genk or at the rehabilitation unit at Sint-Barbara, Lanaken and Cliniques Saint-Luc with medical services on site. All participants will be monitored for fatigue and pain pre, during and at post-intervention daily. The researchers (PI of project [Dr Peter Hallet, ZOL] Postdoctoral Researcher [Dr Lisa Tedesco Triccas, UHasselt] and PhD/Masters Students [UHasselt) will conduct the clinical tests and will conduct the rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

1. a first-ever unilateral, diagnosed stroke by a neurologist as defined by the World Health Organisation,
2. been admitted to the acute hospital for rehabilitation,
3. UL hemiparesis or hemiplegia with a ≥ trace of muscle contraction (≥grade 1 at wrist extensors measured by the MRC Scale and severely motor affected by score of 2 or 3 on item number 5 on the NIH Stroke Scale (NIHSS),
4. the age of > 18 years and (e) the ability to provide informed consent.

Exclusion Criteria:

1. other neurological impairments that could interfere with the protocol such as multiple sclerosis and Parkinson's
2. serious communication, cognitive and language deficits which might hamper the assessment (score of >1 on the command item of the NIHSS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of Motor Recovery after Stroke | baseline
  a stroke-specific, performance-based impairment index.The scale is comprised of five domains and there are 155 items in total (motor functioning, sensory functioning, balance, joint range motion, joint pain). Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.
Fugl-Meyer Assessment of Motor Recovery after Stroke | day 6
  a stroke-specific, performance-based impairment index.The scale is comprised of five domains and there are 155 items in total (motor functioning, sensory functioning, balance, joint range motion, joint pain). Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.
Fugl-Meyer Assessment of Motor Recovery after Stroke | day 9
  a stroke-specific, performance-based impairment index.The scale is comprised of five domains and there are 155 items in total (motor functioning, sensory functioning, balance, joint range motion, joint pain). Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.
Fugl-Meyer Assessment of Motor Recovery after Stroke | day 12
  a stroke-specific, performance-based impairment index.The scale is comprised of five domains and there are 155 items in total (motor functioning, sensory functioning, balance, joint range motion, joint pain). Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.
Fugl-Meyer Assessment of Motor Recovery after Stroke | day 15
  a stroke-specific, performance-based impairment index.The scale is comprised of five domains and there are 155 items in total (motor functioning, sensory functioning, balance, joint range motion, joint pain). Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.

SECONDARY OUTCOMES:
Motricity index | day 3
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 4
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 5
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 6
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 7
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 8
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 9
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 10
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 11
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 12
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 13
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 14
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Motricity index | day 15
  Measurement of upper limb strength. The weighted score based on the ordinal 6 point scale of Medical Research Council was used to measure maximal isometric muscle strength.
Visual Analog Scale of Fatigue (VAS-f) | day 3
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 4
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 5
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 6
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 7
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 8
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 9
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 10
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 11
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 12
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 13
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 14
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Visual Analog Scale of Fatigue (VAS-f) | day 15
  The scale consists of 18 items relating to the subjective experience of fatigue.Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10).
Borg RPE Scale | day 3
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 4
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 5
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 6
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 7
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 8
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 9
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 10
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 11
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 12
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 13
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 14
  Measurement of physical activity intensity (6 to 20 scale)
Borg RPE Scale | day 15
  Measurement of physical activity intensity (6 to 20 scale)
Numeric rating scale pain | day 3
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 4
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 5
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 6
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 7
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 8
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 9
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 10
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 11
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 12
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 13
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 14
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Numeric rating scale pain | day 15
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, prof. dr., Principal Investigator — Hasselt University; Lisa Tabone, dr., Study Chair — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

REFERENCES:
- [Derived] Triccas LT, Hallet P, Cardeynaels S, Ward N, Bertels N, Thijs L, Lejeune T, Lamers I, Spooren A, Feys P. Higher Doses of Intensive Upper Limb Rehabilitation for Moderate to Severe Impairment in Acute, Subacute Stroke: Phase I Dose Escalation Study. Neurorehabil Neural Repair. 2025 Sep;39(9):752-764. doi: 10.1177/15459683251338797. Epub 2025 Jun 28. PMID 40579997